CLINICAL TRIAL: NCT00906191
Title: An Open-Label, Single-Dose, Nonrandomized Study Of The Mass Balance And Metabolic Disposition Of Orally Administered 14C-Labeled SAM-531 In Healthy Male Subjects
Brief Title: Study Evaluating How Quickly And To What Extent The 14-Carbon-SAM-531 Is Absorbed/Converted/Eliminated In Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3193A1-1114
Record Dates: First submitted 2009-05-11; First posted 2009-05-21 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Single oral dose
  Interventions: Drug: SAM-531

INTERVENTIONS:
Drug: SAM-531

SUMMARY:
The objective of this study is to investigate how quickly and to what extent the 14-Carbon labeled SAM-531 is absorbed into the bloodstream, converted and eliminated from the body after oral administration in healthy male subjects. As 14-Carbon labeled SAM-531 is radioactive, this enables the compound to be traced in blood, urine and feces.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 50 years inclusive at screening
* Healthy as determined by the investigator on the basis of screening evaluations

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Radioactivity measurements in blood, urine and feces and pharmacokinetic parameters (Cmax, AUC, terminal elimination half life, total clearance and volume of distribution in the plasma ; urine clearance ; metabolite profiling in plasma, urine and feces.) | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Zuidlaren, Netherlands